CLINICAL TRIAL: NCT01091298
Title: Phase I Randomized Double-blind Placebo-controlled Study to Evaluate the Safety and Tolerability of a Single Administration (10e6.25 FFU of Each Constituent Serotype Per 0.5 ml) of Live Attenuated Tetravalent (G1-G4) Bovine-human Reassortant Rotavirus Vaccine [BRV-TV] Administered to Healthy Indian Adult Males
Brief Title: A Study to Evaluate the Safety of Tetravalent Rotavirus Vaccine in Healthy Indian Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: Head- Research and Development, Shantha Biotechnics Limited
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SBL/BRVTV/Form1/Adlts/PhI/2010
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Safety of vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine (BRV-TV)
- Group 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine (BRV-TV) — Single dose (0.5 mL) of the vaccine administered orally
  Arms: Group 1
Other: Placebo — Single dose (0.5 mL) of the placebo administered orally
  Arms: Group 2

SUMMARY:
This is a Phase I study to evaluate the safety and tolerability of the tetravalent rota virus vaccine in healthy Indian adult male volunteers administered a single dose of the vaccine at the highest possible viral concentration in 0.5 mL of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Indian adult male volunteers.
* No apparent signs or symptoms of ill health.
* Properly informed about the study and having signed the informed consent form (ICF). In case of the volunteer being unable to read or write, having had the ICF explained to them in the presence of a study independent witness and the witness having signed the ICF;
* Subject available for the entire period of the study and reachable by study staff for post-vaccination follow-up.

Exclusion Criteria:

* Known or suspected impairment of immunological function;
* Known hypersensitivity to any component of the rotavirus vaccine;
* Fever, with axillary temperature ≥38.1oC (≥100.5oF); measured by study staff.
* History of chronic diarrhea;
* Clinical evidence of active gastrointestinal illness;
* Receipt of any intramuscular (IM), oral, or intravenous (IV) corticosteroid treatment in the past 30 days
* Subjects suspected to be HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) positive from the available clinical history
* Prior receipt of a blood transfusion or blood products, including immunoglobulins;
* Any subject who cannot be adequately followed for safety;
* Any conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Subject unable to maintain diary card

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Severity and causality of all Adverse Events following the dose of vaccine/placebo | upto 10 days following administration of vaccine/placebo
  The frequency, severity and causality of all solicited and unsolicited adverse events following administration of a single dose of the vaccine as compared to placebo

SECONDARY OUTCOMES:
The frequency and the percentage change, as compared to baseline, in the protocol defined laboratory parameters following the single dose of Vaccine/placebo | Upto 10 days following administration of vaccine/placebo
  The frequency, percentage change, as compared to baseline, and causality of all the defined laboratory parameters following administration of a single dose of the vaccine as compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India